CLINICAL TRIAL: NCT00704574
Title: Safety of Levemir® (Insulin Detemir) Treatment in Children and Adolescents With Type 1 Diabetes (PREDICTIVE™ - Youth)
Brief Title: Observational Study to Observe the Safety of Levemir® Treatment in Children and Adolescents With Type 1 Diabetes
Acronym: PREDICTIVE™
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-1920
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — No extra intervention, only normal clinical practise for treatment of type 1 diabetes
  Other Names: Levemir®

SUMMARY:
This observational study is conducted in Europe. The trial aims to observe the incidence of serious adverse drug reactions in children and adolescents with type 1 diabetes during Levemir® treatment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained prior to any trial-related activities
* Any patient with diabetes type 1 is eligible for the study, including newly
* The selection of the patients will be at the discretion of the individual physician

Exclusion Criteria:

* Type 2 diabetes
* Currently treated with Levemir®

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children Age 6 - 18 with type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse drug reactions, including major hypoglycaemic events | after 6 month treatment

SECONDARY OUTCOMES:
Number of all hypoglycaemic events | after 6 month treatment
Number of adverse drug reactions | after 6 month treatment
BMI changes | after 6 month treatment
HbA1c | after 6 month treatment
Variability in FPG (Fasting Plasma Glucose) | after 6 month treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Lund, Sweden

REFERENCES:
- [Result] Carlsson A, Forsander G, Ludvigsson J, Larsen S, Ortqvist E; Swedish PREDICTIVE-Youth Study Group. A multicenter observational safety study in Swedish children and adolescents using insulin detemir for the treatment of type 1 diabetes. Pediatr Diabetes. 2013 Aug;14(5):358-65. doi: 10.1111/pedi.12019. Epub 2013 Mar 1. PMID 23448369
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com